CLINICAL TRIAL: NCT01968980
Title: A 52 Week, Phase 3 Double-blind, Randomized, Placebo-controlled, Parallel-group Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 In Subjects With Heterozygous Familial Hypercholesterolemia
Brief Title: A 52 Week Study To Assess The Use Of Bococizumab (PF-04950615; RN316) In Subjects With Heterozygous Familial Hypercholesterolemia
Acronym: SPIRE-FH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1481021; 2013-002644-87 (EudraCT Number); SPIRE-HF (Other: Alias Study Number)
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: High Risk of cardiovascular events; Heterozygous familial hypercholesterolemia
MeSH Terms: interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bococizumab (PF-04950615;RN316) (Experimental): Bococizumab (PF-04950615;RN316)
  Interventions: Drug: Bococizumab (PF-04950615;RN316)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bococizumab (PF-04950615;RN316) — 150 mg every 2 weeks, subcutaneous injection, 12 months
  Arms: Bococizumab (PF-04950615;RN316)
Other: Placebo — subcutaneous injection every 2 weeks for 12 months
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized study in subjects with heterozygous familial hypercholesterolemia receiving highly effective statins to assess the safety, efficacy and tolerability of Bococizumab (PF-04950615; RN316) to lower LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a statin.
* Fasting LDL-C > 70 mg/dL and triglyceride <=400 mg/dL.
* High or very high risk of incurring a cardiovascular event.
* Heterozygous familial hypercholesterolemia.

Exclusion Criteria:

* Pregnant or breastfeeding females.
* Cardiovascular or cerebrovascular event of procedures during the past 30 days.
* Congestive heart failure NYHA class IV.
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (88):
- United States (22):
  - IMD Medical Group, Los Angeles, California
  - Hartford Hospital, JB704, Hartford, Connecticut
  - Best Quality Research, Inc., Hialeah, Florida
  - Medical Research Center, Miami, Florida
  - Premier Research Associate, Inc, Miami, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - NewPhase Clinical Trials, Corp., Miami Beach, Florida
  - Om Medical, Las Vegas, Nevada
  - The University of North Carolina at Chapel Hill Center for Heart & Vascular Care, Chapel Hill, North Carolina
  - The University of North Carolina Hospitals - Clinical and Translational Research Center Clinic, Chapel Hill, North Carolina
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Oklahoma Heart Hospital Physicians, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - OnSite Clinical Solutions, LLC, Gaffney, South Carolina
  - Galenos Research, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - Focus Clinical Research, LLC, Draper, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
- Bulgaria (4):
  - SHAT in Cardiology EAD, Pleven
  - UMHAT "Sveti Georgi" EAD, Clinic of Cardiology, Plovdiv
  - Second MHAT - Sofia EAD, Sofia
  - MHAT "Sveta Anna", Clinic of Internal Diseases, Sofia
- Canada (9):
  - St. Paul's Hospital, Healthy Heart, Vancouver, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - Asper Clinical Research Institute, Winnipeg, Manitoba
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut de Recherches Cliniques de Montreal, Montreal, Quebec
  - Clinique des maladies lipidiques de Quebec Inc, Québec, Quebec
- Finland (6):
  - Helsinki Central University Hospital, Helsinki
  - Pohjois-Karjala Projekti Saatio/Ita-Suomen, Joensuu
  - Pohjois-Karjala Projekti Saatio, Joensuu
  - Laakarikeskus Aava Kerava/Aava Kerava Medical Center, Kerava
  - Oulu University Hospital, Oulu
  - Division of Medicine Turku University Hospital, Turku
- Italy (4):
  - Policlinico "Paolo Giaccone", Palermo, PA
  - Ospedale "Santa Maria della Misericordia", Perugia, PG
  - Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Azienda Ospedaliero Universitaria "Federico II" di Napoli, Napoli
- Netherlands (9):
  - St. Franciscus Gasthuis, Rotterdam, South Holland
  - Admiraal de Ruyter ziekenhuis, Goes, Zeeland
  - Academic Medical Center, Amsterdam
  - Amphia Hospital, Breda
  - Deventer Ziekenhuis, Deventer
  - Rotterdam Research Institute, Rotterdam
  - Albert Schweitzer Hospital, Sliedrecht
  - Hagaziekenhuis, The Hague
  - UMC Utrecht, Utrecht
- Norway (2):
  - Oslo Universitetssykehus HF, Oslo
  - Oslo Universitetssykehus HF, Ulleval, Oslo
- Poland (3):
  - NZOZ Vitamed, Bydgoszcz
  - NZOZ Centrum Zdrowia i Profilaktyki Dabie Sp zo.o., Krakow
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek Henryk Rudzki S.C, Ruda Śląska
- South Africa (11):
  - IATROS International, Bloemfontein, Free State
  - Unitas hospital, Centurion, Gauteng
  - Midrand Medical Centre, Halfway House, Gauteng
  - Medipark Centre for Clinical Research, Pretoria, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Chelmsford Medical Centre 3, Durban, KwaZulu-Natal
  - Tiervlei Trial Centre, Karl Bremer Hospital, Bellville, Cape Town, Western Cape
  - TREAD Research cc., Parow, Cape Town, Western Cape
  - Synexus Helderberg Clinical Research Centre, Somerset West, Western Cape
- Spain (10):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico Universitario, Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Fundacion Jimenez Diaz; Servicio de Medicina Interna, Madrid
  - Hospital Clinico San Carlos; U. de Lipidos; Medicina Interna III, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario Miguel Servet; Medicina Interna, Zaragoza
- United Kingdom (8):
  - Clinical Trials Pharmacy, 4th Floor Inpatient Pharmacy, Manchester, Greater Manchester
  - Pennine Acute Hospitals NHS Trust, Oldham, Greater Manchester
  - East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire
  - Burton Hospitals NHS Foundation Trust, Burton-on-Trent, Staffordshire
  - Heart of England NHS Foundation Trust, Birmingham, West Midlands
  - Royal Free London NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Peterborough and Stamford Hospitals NHS Foundation Trust, Peterborough

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] McCush F, Wang E, Yunis C, Schwartz P, Baltrukonis D. Anti-drug Antibody Magnitude and Clinical Relevance Using Signal to Noise (S/N): Bococizumab Case Study. AAPS J. 2023 Sep 2;25(5):85. doi: 10.1208/s12248-023-00846-x. PMID 37658997
- [Derived] Chasman DI, Hyde CL, Giulianini F, Danning RD, Wang EQ, Hickling T, Ridker PM, Loomis AK. Genome-wide pharmacogenetics of anti-drug antibody response to bococizumab highlights key residues in HLA DRB1 and DQB1. Sci Rep. 2022 Mar 11;12(1):4266. doi: 10.1038/s41598-022-07997-5. PMID 35277540
- [Derived] Ridker PM, Rose LM, Kastelein JJP, Santos RD, Wei C, Revkin J, Yunis C, Tardif JC, Shear CL; Studies of PCSK9 Inhibition and the Reduction of vascular Events (SPIRE) Investigators. Cardiovascular event reduction with PCSK9 inhibition among 1578 patients with familial hypercholesterolemia: Results from the SPIRE randomized trials of bococizumab. J Clin Lipidol. 2018 Jul-Aug;12(4):958-965. doi: 10.1016/j.jacl.2018.03.088. Epub 2018 Apr 3. PMID 29685591
- [Derived] Ridker PM, Tardif JC, Amarenco P, Duggan W, Glynn RJ, Jukema JW, Kastelein JJP, Kim AM, Koenig W, Nissen S, Revkin J, Rose LM, Santos RD, Schwartz PF, Shear CL, Yunis C; SPIRE Investigators. Lipid-Reduction Variability and Antidrug-Antibody Formation with Bococizumab. N Engl J Med. 2017 Apr 20;376(16):1517-1526. doi: 10.1056/NEJMoa1614062. Epub 2017 Mar 17. PMID 28304227
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481021&StudyName=A%2052%20Week%20Study%20To%20Assess%20The%20Use%20Of%20RN316%20%28PF-04950615%29%20In%20Subjects%20With%20Heterozygous%20Familial%20Hypercholesterolemia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to PF-04950615 subcutaneous (SC) injection once in every 2 weeks over a period of 52 weeks. Participants were followed up to 58 weeks.
- PF--04950615: Participants received PF-04950615 150 milligram (mg) SC injection once in every 2 weeks over a period of 52 weeks. Participants were followed up to 58 weeks.
Period: Overall Study
Arm/Group | Placebo | PF--04950615
Started | 185 | 185
Completed | 169 | 171
Not Completed | 16 | 14
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 3
Not completed — Does not meet entry criteria | 1 | 3
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Other unspecified | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF--04950615 | Total
Number analyzed (Participants) | 185 | 185 | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.2) | 56.5 (10.5) | 56.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 73 | 155
  Male | 103 | 112 | 215

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 175 | 166
percent change | -0.3 (18.30) | -54.2 (29.34)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; LS-mean difference,associated 95 percent (%) confidence intervals (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures (MMRM); Least square (LS) mean difference = -54.5, 95% CI 2-sided [-59.5 to -49.5], Standard Error of Mean 2.54

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 175 | 166
percent change | -0.0 (14.45) | -37.0 (19.82)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; LS-mean difference,associated 95% confidence intervals (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -37.6, 95% CI 2-sided [-41.1 to -34.1], Standard Error of Mean 1.77

3. Secondary Outcome: Percent Change From Baseline in Non High Density Lipoprotein Cholesterol (Non HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 175 | 166
percent change | 0.4 (17.89) | -49.9 (26.80)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -51.0, 95% CI 2-sided [-55.7 to -46.4], Standard Error of Mean 2.36

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 175 | 166
percent change | 0.4 (15.96) | -47.5 (28.89)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -48.0, 95% CI 2-sided [-52.8 to -43.2], Standard Error of Mean 2.44

5. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 172 | 166
percent change | 2.2 (27.21) | -26.4 (23.63)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -28.6, 95% CI 2-sided [-33.9 to -23.2], Standard Error of Mean 2.73

6. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 175 | 166
percent change | -0.3 (12.99) | 6.3 (15.11)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = 7.0, 95% CI 2-sided [4.1 to 9.9], Standard Error of Mean 1.47

7. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 24 (n =175, 173) | 2.7 (25.38) | -50.1 (32.94)
  Week 52 (n =169, 171) | 3.5 (21.49) | -45.3 (30.87)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; Week 24: LS-mean difference,associated 95% confidence intervals (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region; Test type: Superiority or Other; LS mean difference = -52.1, 95% CI 2-sided [-58.2 to -46.0], Standard Error of Mean 3.10
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; Week 52: LS-mean difference,associated 95% confidence intervals (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region; Test type: Superiority or Other; LS mean difference = -48.0, 95% CI 2-sided [-53.6 to -42.3], Standard Error of Mean 2.87

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 24 (n =176, 173) | 1.6 (19.10) | -34.4 (21.44)
  Week 52 (n =169, 171) | 1.2 (15.82) | -31.0 (21.50)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -35.8, 95% CI 2-sided [-40.0 to -31.6], Standard Error of Mean 2.12
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -31.8, 95% CI 2-sided [-35.8 to -27.8], Standard Error of Mean 2.02

9. Secondary Outcome: Percent Change From Baseline in Non High Density Lipoprotein Cholesterol (Non HDL-C) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 24 (n =174, 173) | 2.4 (24.06) | -46.7 (29.88)
  Week 52 (n =169, 171) | 1.2 (19.25) | -41.8 (29.99)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -48.5, 95% CI 2-sided [-54.1 to -42.8], Standard Error of Mean 2.86
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -42.2, 95% CI 2-sided [-47.5 to -36.9], Standard Error of Mean 2.71

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 24 (n =176, 171) | 2.6 (19.29) | -44.8 (30.40)
  Week 52 (n =169, 171) | 1.7 (16.45) | -39.3 (28.89)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -46.8, 95% CI 2-sided [-52.1 to -41.6], Standard Error of Mean 2.67
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -40.5, 95% CI 2-sided [-45.5 to -35.5], Standard Error of Mean 2.53

11. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 24 (n =175, 172) | 14.6 (157.93) | -21.2 (48.77)
  Week 52 (n =168, 171) | 1.3 (30.50) | -15.1 (68.22)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -35.1, 95% CI 2-sided [-59.8 to -10.3], Standard Error of Mean 12.58
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -15.3, 95% CI 2-sided [-26.3 to -4.4], Standard Error of Mean 5.58

12. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 24 (n =174, 173) | 0.9 (14.19) | 6.6 (12.85)
  Week 52 (n =169, 171) | 2.2 (14.51) | 4.7 (14.30)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 5.9, 95% CI 2-sided [3.1 to 8.7], Standard Error of Mean 1.42
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 2.9, 95% CI 2-sided [-0.1 to 5.9], Standard Error of Mean 1.53

13. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 12 (n =175, 166) | 7.1 (41.23) | -8.7 (38.07)
  Week 24 (n =176, 173) | 7.6 (51.97) | -9.0 (40.01)
  Week 52 (n =169, 171) | 4.9 (33.03) | -3.4 (58.27)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; Week 12: LS-mean difference,associated 95% confidence intervals (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region; Test type: Superiority or Other; LS Mean Difference = -17.0, 95% CI 2-sided [-25.3 to -8.7], Standard Error of Mean 4.22
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -17.4, 95% CI 2-sided [-27.0 to -7.8], Standard Error of Mean 4.90
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -9.5, 95% CI 2-sided [-19.4 to 0.4], Standard Error of Mean 5.04

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 12 (n =175, 166) | -0.5 (11.70) | 4.8 (12.15)
  Week 24 (n =176, 172) | -0.6 (10.69) | 3.9 (10.72)
  Week 52 (n =169, 171) | 0.3 (12.02) | 3.0 (11.53)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 5.3, 95% CI 2-sided [2.9 to 7.8], Standard Error of Mean 1.25
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 4.6, 95% CI 2-sided [2.5 to 6.8], Standard Error of Mean 1.10
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 3.0, 95% CI 2-sided [0.5 to 5.4], Standard Error of Mean 1.22

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-II (ApoA-II) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 12 (n =175, 166) | -2.6 (13.34) | -1.6 (15.68)
  Week 24 (n =175, 170) | -2.8 (11.88) | -1.8 (13.45)
  Week 52 (n =167, 171) | -3.5 (11.90) | -2.4 (14.50)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.7, 95% CI 2-sided [-2.3 to 3.6], Standard Error of Mean 1.50
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.6, 95% CI 2-sided [-1.9 to 3.2], Standard Error of Mean 1.31
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 0.8, 95% CI 2-sided [-1.9 to 3.6], Standard Error of Mean 1.39

16. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein Cholesterol (VLDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percent change
  Week 12 (n =175, 166) | 7.1 (41.23) | -8.7 (38.07)
  Week 24 (n =176, 173) | 7.6 (51.97) | -9.0 (40.01)
  Week 52 (n =169, 171) | 4.9 (33.03) | -3.4 (58.27)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -17.0, 95% CI 2-sided [-25.3 to -8.7], Standard Error of Mean 4.22
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -17.4, 95% CI 2-sided [-27.0 to -7.8], Standard Error of Mean 4.90
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -9.5, 95% CI 2-sided [-19.4 to 0.4], Standard Error of Mean 5.04

17. Secondary Outcome: Absolute Change From Baseline in Low Density Lipoprotein (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
milligram per deciliter (mg/dL)
  Baseline (n= 185, 185) | 150.0 (59.75) | 144.2 (41.96)
  Change at Week 12 (n= 175, 166) | -3.0 (30.47) | -79.1 (46.97)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -78.8, 95% CI 2-sided [-86.2 to -71.4], Standard Error of Mean 3.75

18. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol (TC) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
mg/dL
  Baseline (n= 185, 185) | 227.2 (67.31) | 220.7 (46.26)
  Change at Week 12 (n= 175, 166) | -2.8 (36.43) | -83.2 (49.51)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -83.2, 95% CI 2-sided [-91.3 to -75.0], Standard Error of Mean 4.15

19. Secondary Outcome: Absolute Change From Baseline in Non- High Density Lipoprotein Cholesterol (Non HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
mg/dL
  Baseline (n= 185, 185) | 178.6 (66.64) | 170.4 (45.12)
  Change at Week 12 (n= 175, 166) | -2.3 (36.24) | -86.0 (51.09)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -87.0, 95% CI 2-sided [-95.4 to -78.7], Standard Error of Mean 4.25

20. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B (ApoB) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
mg/dL
  Baseline (n= 185, 185) | 115.9 (35.25) | 112.8 (26.26)
  Change at Week 12 (n= 175, 166) | -0.9 (20.51) | -53.7 (33.07)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -53.8, 95% CI 2-sided [-59.2 to -48.5], Standard Error of Mean 2.71

21. Secondary Outcome: Absolute Change From Baseline in Lipoprotein (a) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
mg/dL
  Baseline (n= 184, 185) | 58.8 (69.88) | 59.7 (63.38)
  Change at Week 12 (n= 172, 166) | -1.4 (14.02) | -14.0 (17.91)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -11.8, 95% CI 2-sided [-14.7 to -8.9], Standard Error of Mean 1.47

22. Secondary Outcome: Absolute Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
mg/dL
  Baseline (n= 185, 185) | 48.6 (11.84) | 50.3 (11.40)
  Change at Week 12 (n= 175, 166) | -0.6 (6.31) | 2.8 (7.89)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 3.5, 95% CI 2-sided [2.0 to 4.9], Standard Error of Mean 0.75

23. Secondary Outcome: Absolute Change From Baseline in Ratio of Total Cholesterol to High Density Lipoprotein Cholesterol (TC/HDL-C Ratio) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
ratio
  Baseline (n =185, 185) | 4.9 (1.81) | 4.6 (1.32)
  Change at Week 12 (n =175, 166) | 0.0 (1.00) | -1.8 (1.29)
  Change at Week 24 (n =174, 173) | 0.0 (1.20) | -1.7 (1.29)
  Change at Week 52 (n =169, 171) | -0.0 (1.00) | -1.5 (1.35)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -2.0, 95% CI 2-sided [-2.2 to -1.8], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -1.8, 95% CI 2-sided [-2.1 to -1.6], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -1.6, 95% CI 2-sided [-1.8 to -1.3], Standard Error of Mean 0.12

24. Secondary Outcome: Absolute Change From Baseline in Ratio of Apolipoprotein B to Apolipoprotein A-I (ApoB/ApoA-I Ratio) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
ratio
  Baseline (n =185, 185) | 0.8 (0.31) | 0.8 (0.23)
  Change at Week 12 (n =175, 166) | 0.0 (0.18) | -0.4 (0.25)
  Change at Week 24 (n =176, 171) | 0.0 (0.17) | -0.4 (0.25)
  Change at Week 52 (n =169, 171) | 0.0 (0.17) | -0.3 (0.25)
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.4, 95% CI 2-sided [-0.5 to -0.4], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; Week 24:LS-mean difference,associated 95% confidence intervals (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region; Test type: Superiority or Other; LS Mean Difference = -0.4, 95% CI 2-sided [-0.4 to -0.4], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; LS Mean Difference = -0.3, 95% CI 2-sided [-0.4 to -0.3], Standard Error of Mean 0.02

25. Secondary Outcome: Percentage of Participants Achieving Low Density Lipoprotein Cholesterol (LDL-C) Level Less Than or Equal to (<=) 100 Milligram Per Deciliter (2.59 Millimoles Per Liter) at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percentage of participants
  Week 12 (n =175, 166) | 13.1 | 83.1
  Week 24 (n =175, 173) | 13.1 | 80.9
  Week 52 (n =169, 171) | 16.6 | 70.8
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; Week 12: Odds ratio, associated 95% confidence interval and p-value from a Logistic Regression Model with fixed effects for treatment group,baseline value and geographical region was used for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 51.8, 95% CI 2-sided [25.24 to 106.10]
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; Week 24: Odds ratio, associated 95% confidence interval and p-value from a Logistic Regression Model with fixed effects for treatment group,baseline value and geographical region was used for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 66.9, 95% CI 2-sided [30.32 to 147.43]
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; Week 52: Odds ratio, associated 95% confidence interval and p-value from a Logistic Regression Model with fixed effects for treatment group,baseline value and geographical region was used for analysis; Test type: Superiority or Other; Odds Ratio (OR) = 22.8, 95% CI 2-sided [11.85 to 44.01]

26. Secondary Outcome: Percentage of Participants Achieving Low Density Lipoprotein Cholesterol (LDL-C) Level Less Than or Equal to (<=) 70 Milligram Per Deciliter (1.81 Millimoles Per Liter) at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
percentage of participants
  Week 12 (n =175, 166) | 1.1 | 66.3
  Week 24 (n =175, 173) | 1.1 | 60.7
  Week 52 (n =169, 171) | 0.6 | 53.2
Statistical Analysis 1: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 25, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 200.8, 95% CI 2-sided [47.16 to 854.60]
Statistical Analysis 2: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 25, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 228.0, 95% CI 2-sided [51.95 to 1000.39]
Statistical Analysis 3: Comparison: Placebo vs PF--04950615; [analysis description as in outcome 25, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 259.9, 95% CI 2-sided [34.87 to 1937.06]

27. Secondary Outcome: Plasma PF-04950615 Concentrations at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: Analysis was performed on all participants who received at least 1 dose of PF-04950615. Here, 'n' signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | PF--04950615
Number analyzed (Participants) | 185
microgram per milliliter
  Week 12 (n =163) | 6.23 (5.657)
  Week 24 (n =167) | 7.00 (6.351)
  Week 52 (n =171) | 4.84 (5.384)

28. Secondary Outcome: Number of Participants With Adverse Events Related to Type 1 or 3 Hypersensitivity Reactions and Injection Site Reactions
Description: Type 1 hypersensitivity or allergic reactions were possible in response to any injected protein and included shortness of breath, urticaria, anaphylaxis and angioedema. Type 3 hypersensitivity reactions were similar to Type 1 hypersensitivity reactions but were likely to be delayed from the time of injection and included symptoms such as rash, urticaria, polyarthritis, myalgia, polysynovitis, fever and if severe then included glomerulonephritis as well. Injection site reaction is a reaction at the site of the subcutaneous injection and characterized by the symptoms of erythema, swelling, tenderness and warmth. Participants with any of the above type 1 or type 3 hypersensitivity reactions and participants with any of the above injection site reactions were reported in this outcome measure.
Time Frame: Baseline up to the end of study (up to 58 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF--04950615
Number analyzed (Participants) | 185 | 185
participants
  With Type 1 or 3 hypersensitivity reactions | 0 | 0
  With Injection site reactions | 1 | 38

29. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb)
Description: Percentage of participants with at least 1 positive ADA titer or 1 positive nAb titer were reported in this outcome measure. ADA titer greater than or equal to (>=) 6.23 were considered as ADA positive and nAb titer level >=1.58 were considered as nAb positive.
Time Frame: Baseline up to the end of study (up to 58 weeks)
Population: Analysis was performed on all participants who received at least 1 dose of PF-04950615.
Measure: Number; unit: percentage of participants
Arm/Group | PF--04950615
Number analyzed (Participants) | 185
percentage of participants
  With positive ADA | 49.7
  With positive nAb | 33

ADVERSE EVENTS:
Time Frame: Baseline up to the end of study (up to 58 weeks)
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Placebo | PF--04950615
Serious Adverse Events (participants affected / at risk) | 22/185 | 24/185
Other Adverse Events (participants affected / at risk) | 36/185 | 70/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=185) | PF--04950615 (N=185)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 3 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Vascular stent restenosis (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/103 | 1/112 — This is gender specific event. The number of participants evaluable for this event are 103 and 112.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Device breakage (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=185) | PF--04950615 (N=185)
Injection site reaction (General disorders) | 1 | 38
Influenza (Infections and infestations) | 6 | 10
Nasopharyngitis (Infections and infestations) | 15 | 15
Upper respiratory tract infection (Infections and infestations) | 7 | 11
Headache (Nervous system disorders) | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.